CLINICAL TRIAL: NCT02416895
Title: Vitamin D Status and in Vivo Immune Function
Brief Title: Vitamin D Status and Immune Function
Status: Completed | Type: Observational
Sponsor: Bangor University (Other)
Collaborators: University of East Anglia (Other)
Responsible Party: Sponsor
Other Study IDs: 165/Gen/10
Record Dates: First submitted 2015-03-25; First posted 2015-04-15 (Estimated); Last update posted 2017-04-05 (Actual); Status verified 2017-03

CONDITIONS: Vitamin D Deficiency
MeSH Terms: conditions — Vitamin D Deficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood serum collected at Week 1 (start of training) and Week 13 (end of training).
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Army recruits: Army recruits at the start of basic training will complete an in vivo immunity model
  Interventions: Other: In vivo immunity model

INTERVENTIONS:
Other: In vivo immunity model — A measure of in vivo immune function.

SUMMARY:
The purpose of this study is to examine the relationship between Vitamin D status and immunity.

DETAILED DESCRIPTION:
Vitamin D is mainly obtained from the sun and follows a seasonal pattern, with Vitamin D levels peaking in summer and reaching a trough during winter. Vitamin D deficiency is associated with impaired immunity. However, knowledge of Vitamin D deficiency with in vivo immunity is limited. This observational study aims to investigate the relationship between Vitamin D status and the in vivo immunity.

ELIGIBILITY:
Inclusion Criteria:

* Passed medical assessment by medical doctor
* Passed audio test (this is part of medical assessment)
* Met physical fitness requirements

Exclusion Criteria:

• Medically deferred by medical doctor

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Young adults who are starting basic training in the army.
Sampling Method: Non-Probability Sample
Enrollment: 264 (Actual)
Dates: Start 2014-04; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Vitamin D measured by liquid chromatography tandem mass spectroscopy | Up to 20 months
  Circulating 25-hydroxy-vitamin D

SECONDARY OUTCOMES:
Immune function measured by analytic biochemistry assay | Up to 20 months
  In vivo immune measure

CONTACTS AND LOCATIONS:
Overall Officials: Julie Greeves, PhD, Principal Investigator — HQ Army Research and Training Division
Locations (1):
- Infantry Training Centre, Catterick, North Yorkshire, United Kingdom

REFERENCES:
- [Derived] Kashi DS, Oliver SJ, Wentz LM, Roberts R, Carswell AT, Tang JCY, Jackson S, Izard RM, Allan D, Rhodes LE, Fraser WD, Greeves JP, Walsh NP. Vitamin D and the hepatitis B vaccine response: a prospective cohort study and a randomized, placebo-controlled oral vitamin D3 and simulated sunlight supplementation trial in healthy adults. Eur J Nutr. 2021 Feb;60(1):475-491. doi: 10.1007/s00394-020-02261-w. Epub 2020 May 10. PMID 32390123
- [Derived] Tang JCY, Jackson S, Walsh NP, Greeves J, Fraser WD; Bioanalytical Facility team. The dynamic relationships between the active and catabolic vitamin D metabolites, their ratios, and associations with PTH. Sci Rep. 2019 May 6;9(1):6974. doi: 10.1038/s41598-019-43462-6. PMID 31061425